CLINICAL TRIAL: NCT05436405
Title: Trans-pedal Access for Endovascular Revascularization in Complex Infra-popliteal Lesions in Critically Ischemic Limb
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: mansouravascular
Record Dates: First submitted 2022-06-15; First posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Critical Lower Limb Ischemia
Keywords: transpedal access; retrogradeangioplasty; critical limb ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- transpedal access (Experimental): Trans-pedal Access for Endovascular Revascularization in patients with failed antegrade access forComplex Infra-popliteal Lesions in Critically Ischemic Limb
  Interventions: Procedure: Trans-pedal access for endovascular revascularization in complex infra-popliteal lesions in critically ischemic limb

INTERVENTIONS:
Procedure: Trans-pedal access for endovascular revascularization in complex infra-popliteal lesions in critically ischemic limb — Briefly, conventional femoral access will be conducted in the traditional manner and involve the sheath while the catheter was introduced close to the proximal degree of lesion.
  Access to a pedal vessel: Using a 21-guage needle or by utilizing a micro puncture access set. Such vessel is recognized using the US probe. such approach performed in 54 patients.a fluoroscopy might enable a good possibility for efficient access. In addition, it was suggested to utilize micro-puncture needle supposed to have echogenic pattern as the tip of regular needle is very hard to visualize utilizing the duplex US probe. Also, use of straight fluoroscopy or road mapping may offer a better chance for successful access, this method is done in 31 cases . Another method is open method (cut down) on tibial vessels, this method is done in 11 cases.

SUMMARY:
Background: critical limb ischemia is one of the most challenging cases we face nowadays with high risk for amputation, retrograde trans-pedal angioplasty offers an alternative technique after failure of traditional ante-grade angioplasty.

Patients and Methods: 96 patients underwent trans-pedal or trans-tibial retrograde angioplasty after failure of the traditional ante-grade angioplasty with the aid of US, 21-gauge needle and 0.018 wire through sheath-less approach as a last chance for revascularization

DETAILED DESCRIPTION:
Study Design: This prospective non randomized study that had been performed at vascular surgery department at Mansoura University Hospital between March 2018 and April 2020, who was selected for 96patients undergoing endovascular BTK revascularization for CLI owing to tibial vascular diseases and gave written informed consent. Such cases who not give good response following traditional ante-grade ipsilateral trans-femoral approach and consequently underwent retrograde Trans-pedal or transtibial access to provide endovascular management for the lesions.

Inclusion criteria:

* all patients aged from (18-80) years, males and female
* patients with 1ry lesion (without previous trial of angioplasty or bypass)
* 2ry lesion (after previous trial of angioplasty or bypass),
* the patients with fountain classification (stage IIB, stage III, stage IV)
* patients with Rutherford classification (grade I "category 3", grade II, Category 4", grade III, Category 4&category 5.

Exclusion criteria:

* patients with untreated osteomyelitis,
* patients with mixed lesions with other comorbidities (CVI & Lymphoedema),
* patients with vasculitis or Buerger's dis.
* Also, who can't give consent (mentally retarded patients) or those with behavioral disorders .

Study tools History Data: included patient's demographics, underlying medical conditions, any previous surgery, transplanted kidney and other associated morbidity.

Examination: Full arterial assessments included pulse examination, and the ABPI (ankle brachial pressure index).

Laboratory: Blood picture, Blood sugar level, Kidney functions, Liver functions and Coagulation profile.

Imaging: Duplex ultra-sonographic (US) examination and CTA. Technique: Entire cases underwent full therapeutic medication prior to interference. Entire cases were tried ante-grade re-vascularization with a subsequent failure. A lower limb angiogram was be ready in entire cases prior to the retrograde procedure performance. Briefly, conventional femoral access will be conducted in the traditional manner and involve the sheath while the catheter was introduced close to the proximal degree of lesion.

Access to a pedal vessel: Using a 21-guage needle with insertion of 0.018-inch wire by sheathless technique (Figure 1) or by utilizing a micro puncture access set. A duplex-guided access has a great importance in terms of evaluation of the pedal as well as tibial blood vessels. Such vessel is recognized using the US probe. Color flow is utilized for identification of the objective artery flow, after that color disappeared while the needle is utilized for accessing the anterior vascular surface by utilizing duplex US , such approach performed in 54 patients. There are technical points worth mentioning utilizing such procedure: usage the smallest ready US as the major ones are bulky and may have a role in interference with the access process. In addition, marked vascular calcification may induce marked shadow making the identification very hard to be detected. In such conditions, a fluoroscopy might enable a good possibility for efficient access. In addition, it was suggested to utilize micro-puncture needle supposed to have echogenic pattern as the tip of regular needle is very hard to visualize utilizing the duplex US probe. Also, use of straight fluoroscopy or road mapping may offer a better chance for successful access, as we mentioned before, this method is done in 31 cases . Appropriate section of the actual place of vascular access is essential for the successfulness of such procedure. Generally, a patent vascular is selected to be the access situation. A micro-puncture needle is utilized for access. Occasionally, bending the needle tip has the ability to make the possibility of vascular evaluation easy which has great importance if the access point in the ATA beyond the ankle. Another method is open method (cut down) on tibial vessels, this method is done in 11 cases. Following evaluating the artery, established by back hemorrhage, the micro puncture access wire is introduced via the needle into the vessels underneath fluoroscopic guide in a retrograde fashion. The needle is removed and micro puncture set (4F) or the balloon itself is passed over the wire to secure the access. According to micro puncture introducer set it includes a 21- gauge, 7- cm echogenic needle, 10 - cm long micro puncture 4-french introducer and 2.9F inner caliber permitting passage of the equipment. When the retrograde introducers are in position, the case is completely heparinized to prevent any thrombus development throughout the interference process. An exchange dimension 0.018-inch wire was utilized to try passing across the disorder in a retrograde manner, it has very accurate outcomes crossing the obstruction for combination of a small sufficient diameter with adequate body support to permit crossing of the obstruction calcified in several patients. The V18 TM Control Wire Guide Wire is specifically beneficial at such condition. It has a hydrophilic tip which may assist in sliding via the blockade with mild frictions, and simultaneously the wire has sufficient stiffness to pass across the overall occlusion. In sometimes, the usage of the 0.018 system only aiming for crossing isn't sufficient. Such condition specifically develops when there are prolonged occlusions and when there is marked calcification. In such patients, additional reinforcement is required for the platform to permit the crossing. Thus, up-sizing to a 0.035 system might help in disorder crossing. When we pass through the disorder, an angiogram from below is conducted to prove the situation in the actual lumen beyond the disorder. The 0.018-inch system and wire were removed and hemostasis secured via digital compression for 8 minutes or by ante-grade balloon dilatation at the site of puncture for about 2-3 minutes.

Patient follow-up: Patients had been evaluated through the ABPI and duplex US examination: immediately, three mo., 6 mo., and 1 year following the surgery.

ELIGIBILITY:
Inclusion Criteria:

* all patients aged from (18-80) years, males and female
* patients with 1ry lesion (without previous trial of angioplasty or bypass)
* 2ry lesion (after previous trial of angioplasty or bypass),
* the patients with fountain classification (stage IIB, stage III, stage IV)
* patients with Rutherford classification (grade I "category 3", grade II, Category 4", grade III, Category 4&category 5.

Exclusion criteria:

* patients with untreated osteomyelitis,
* patients with mixed lesions with other comorbidities (CVI & Lymphoedema),
* patients with vasculitis or Buerger's dis.
* Also, who can't give consent (mentally retarded patients) or those with behavioral disorders .

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
primary patency | one year
  patency of the vessels after intervention
amputation free survival rates | one year
  limb salvage after precedure
30 days' mortality and morbidity. | 30 days
  major adverse effects related to procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No